CLINICAL TRIAL: NCT00412399
Title: Job Adaptation in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Other Study IDs: 97068
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2006-12-18 (Estimated); Status verified 2006-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Employment; Negative workplace events; Healthy controls; Fatigue; Physical activity
MeSH Terms: conditions — Arthritis, Rheumatoid; Fatigue; Motor Activity

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective

SUMMARY:
The specific aim of this study is to compare the rate of negative work role events in individuals with rheumatoid arthritis compared to healthy controls.

DETAILED DESCRIPTION:
Rheumatoid arthritis can cause multiple socio-medical disabilities, with work disability among the most marked. While a major focus has been documenting the rates of job loss and returning patients to the workforce, there is little information about how to foster job retention in those still employed. The goals of this study are to document negative workplace events over 1 year in 122 employed patients with rheumatoid arthritis, and to compare these to 122 healthy controls, who are included to account for the effects of socioeconomic status on employment. Events will be recorded with the work domain of the Psychiatric Epidemiology Research Life Events Scale. Additional goals are to compared fatigue, physical activity, functional status and sleep disturbances as covariates.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible if they are:

  * over age 18;
  * meet American Rheumatism Association criteria for rheumatoid arthritis; and
  * are employed for salary or monetary reimbursement.
* Controls are eligible if they are:

  * over age 18;
  * have no major comorbidity; and
  * are employed for salary or monetary reimbursement.

Exclusion Criteria:

* Patients and controls are excluded if they:

  * have cognitive deficits and cannot provide informed consent;
  * do not speak English or Spanish; or
  * their physicians do not grant permission to enroll them.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 244
Dates: Start 1999-06; Study Completion 2001-10

CONTACTS AND LOCATIONS:
Overall Officials: Carol A Mancuso, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (2):
- United States (2):
  - Cornell Internal Medicine Associates, New York, New York
  - Hospital for Special Surgery, New York, New York

REFERENCES:
- [Background] Mancuso CA, Paget SA, Charlson ME. Adaptations made by rheumatoid arthritis patients to continue working: a pilot study of workplace challenges and successful adaptations. Arthritis Care Res. 2000 Apr;13(2):89-99. PMID 14635282